CLINICAL TRIAL: NCT05924009
Title: Characterization of Gastric Evoked Potentials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, David Levinthal, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY23030127; R21NS123502 (NIH)
Record Dates: First submitted 2023-06-16; First posted 2023-06-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants
  Interventions: Procedure: Transcranial Magnetic Stimulation, TMS

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation, TMS — The best location for evoking an electromyographic (EMG) response of the first dorsal interosseus (FDI) muscle in the dominant hand and the minimum stimulation intensity required to evoke a certain EMG response amplitude (Motor Threshold, MT) are used as reference to determine the best location and stimulation parameters to evoke GEPs.
  After identification of the GEP hot-spot, a water load test is administered to determine whether satiety shapes GEP responses.
  In subsequent study visits, the water load test is preceded by application of neuromodulatory repetitive TMS (rTMS), targeted to the GEP hotspot.

SUMMARY:
This is an exploratory study that will determine and standardize how best to record gastric evoked potentials (GEPs) elicited by a non-invasive method of brain stimulation (Transcranial Magnetic Stimulation, TMS), by optimizing the TMS parameters and cortical sites necessary to evoke GEPs.

DETAILED DESCRIPTION:
The overall goal of this exploratory study is to determine the optimal conditions to elicit gastric evoked potentials (GEPs) with Transcranial Magnetic Stimulation (TMS).

Aim 1: Determine the optimal stimulation parameters and the optimal location for eliciting GEPs in cortical motor areas.

Aim 2: Determine whether various modes of repetitive TMS (rTMS) neuromodulation targeted to GEP hotspots shape gastric motor responses to a water load.

The investigators will record some clinical, demographic, and autonomic data (i.e. EKG) in our enrolled subjects. Secondary analyses will use these variables as covariates to investigate any systematic impact on the measures from Aims 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* psychosis or altered cognitive status
* history of head injury, metal in the skull, stroke, or a history of seizures, loss of consciousness or syncope
* implantable devices, such as a pacemaker or nerve stimulator
* current use of antiepileptic medications or current use of the following medications or substances which are known to lower the seizure threshold: Clozapine (Clozaril), Chlorpromazine (Thorazine), amphetamines or methamphetamine, Ecstasy, Ketamine, Angel Dust/PCP, cocaine, or 3 or more alcoholic drinks per day
* pregnancy
* BMI > 30
* history of bariatric surgery such as sleeve gastrectomy or Roux-en-Y gastric bypass
* diabetes
* suffering from a neurodegenerative disorder.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 155 (Estimated)
Dates: Start 2023-06-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in GEP hotspot location | Multiple study sessions spanning up to 12 months
  Stimulation location evoking the largest GEP response, relative to FDI hotspot location
Change in optimal stimulation parameters at GEP hotspot | Multiple study sessions spanning up to 12 months
  Stimulation pattern (single pulses or brief bursts) and strength relative to MT for FDI

SECONDARY OUTCOMES:
Effect of satiety | Multiple study sessions spanning up to 12 months
  Change in GEP amplitude after water load test
Effect of neuromodulation | Multiple study sessions spanning up to 12 months
  Change in GEP amplitude when water load test is preceded by rTMS

CONTACTS AND LOCATIONS:
Overall Officials: David J Levinthal, MD PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to place participant data into a open-access, shared data repository. However, a data sharing agreement can be made if requested.